CLINICAL TRIAL: NCT05555277
Title: Retrospective Examination of Electroencephalography Signals of Individuals With Different Eating Disorders
Status: Completed | Type: Observational
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Fatma Demir, Research Assistant, Uskudar University
Other Study IDs: UskudarUni1
Record Dates: First submitted 2022-09-20; First posted 2022-09-26 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa
Keywords: eating disorders; electroencephalography; depression
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa; Feeding and Eating Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anorexia Nervosa: Individuals aged 18 years and younger with anorexia nervosa who have beck depression inventory, beck anxiety inventory, eating attitude test-40 and EEG data in their patient file.
  Interventions: Other: No interventions - retrospective data collection
- Bulimia Nervosa: Individuals aged 18 years and younger with bulimia nervosa who have beck depression inventory, beck anxiety inventory, eating attitude test-40 and EEG data in their patient file.
  Interventions: Other: No interventions - retrospective data collection

INTERVENTIONS:
Other: No interventions - retrospective data collection — The differences between the two diagnoses were investigated by using the scale results and EEG data in the patient files.

SUMMARY:
The aim of this study was to investigate the difference between electroencephalography (EEG) data and current psychological status of individuals diagnosed with anorexia nervosa (AN) and bulimia nervosa (BN).

DETAILED DESCRIPTION:
The data used in this study were obtained from individuals aged 18 and younger with eating disorders who applied to Üsküdar University NP Istanbul Brain Hospital. Two different diagnostic groups, Anorexia Nervosa and Bulimia Nervosa, were included in the study. Demographic information, secondary diagnosis status, Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), Eating Attitude Test - 40 (EAT-40) scores and EEG data were used to investigate the differences between eating disorders. Comparison of neurological differences between individuals with AN and BN was done retrospectively.

This information, which will be obtained for AN and BN, which are diseases in which severe deterioration in behavior and perception are seen, can give advice to experts in planning treatment and rehabilitation processes.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with anorexia nervosa or bulimia nervosa to the DSM-V diagnostic criteria
* 18 years and younger
* Having an EEG data

Exclusion Criteria:

* Having an EEG data taken in a center other than NP Istanbul Brain Hospital
* Lack of "Beck Depression Inventory", "Beck Anxiety Inventory" and "Eating Attitude Test-40" scale values in the patient file

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals aged 18 years or younger with AN and BN who were administered scales of depression, anxiety and eating attitudes
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-26 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Differences between EEG data of patients with anorexia nervosa and bulimia nervosa | April 2022-September 2022
  EEG data of individuals with eating disorders were compared.
Differences between depression levels of patients with anorexia nervosa and bulimia nervosa | April 2022-September 2022
  Depression levels of individuals with eating disorders were compared.
Differences between anxiety levels of patients with anorexia nervosa and bulimia nervosa | April 2022-September 2022
  Anxiety levels of individuals with eating disorders were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Demir, Principal Investigator — Research assistant; Alper Evrensel, Study Chair — Associate professor; Tuğçe Ballı Altuğlu, Study Director — Assistant professor
Locations (1):
- Fatma Demir, Üsküdar, İ̇stanbul, Turkey (Türkiye)